Cell Phone Support to Promote Medication Adherence Among Adolescents and Young Adults With Chronic Illness

NCT04241627

8/8/2022

This randomized pilot trial tested three different digital health interventions against one another (CPS-C, n = 11, CPS-T, n = 12, and ATR, n = 11). We are interested in the impact on self-reported medication adherence. We have 6 different measures of dependent variables (VAS1w, VAS2w, VAS3w, VAS1m, VAS2m, VAS3m). We assessed our dependent variables 4 occasions, at 0 weeks (pre-tx), 6 weeks (mid-tx), 12 weeks (post-tx), and 18 weeks (follow-up). We would like to run mixed-effect models to test for intervention effects of 1) both CPS conditions (CPS-C and CPS-T, n = 23) versus ATR (n = 11); and 2) the CPS conditions against each other, ignoring ATR (CPS-C, n = 11 versus CPS-T, n = 12). I also have covariates (sex assigned at birth, diagnosis, age) that we can include during nested model building procedures, and include in final reported models if they lead to best fit.

Can we begin by examining the distributions of our dependent variables, and discuss whether we should use linear mixed-effects models; otherwise, we may need to transform or dichotomize the outcome or use a different type of model (poissson? Negative binomial?) to ensure model assumptions are met?

Then, can we evaluate the impact of missing data on my results by re-running these analyses using inverse probably weighting. It is possible that missing data will not be completely at random (i.e., participants with lower medication adherence may also be less likely to adhere to the online survey schedule).

Finally, I would like to calculate effect sizes for subgroups (see the final table). See tables on the next pages.

## **Blank Tables**

Table 5
Best-Fitting Models Predicting Self-Reported Adherence for Both CPS Conditions (C and T) versus ATR (N = 34)

| Dependent<br>Variables | VAS1 | lw | | VAS2 | VAS2w | | | VAS3w | | | m | VAS2 | 2m | | VAS3m | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variables | E (' ) | CI. | ı | E 4' 4 | CI. | l | E 4: 4 | $\alpha$ | | Г.: . | $\alpha$ | ı | E 4: 4 | - CI | | Г. /· / | - CI | $\overline{1}$ |
| | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p |
| Fixed Effects | | | | | | | | | | | | | | | | | | |
| Intercept | | | | | | | | | | | | | | | | | | |
| Time | | | | | | | | | | | | | | | | | | |
| Intervention | | | | | | | | | | | | | | | | | | |
| Group (both CPS | | | | | | | | | | | | | | | | | | |
| versus ATR) | | | | | | | | | | | | | | | | | | |
| Random Effects | | | | | | | | | | | | | | | | | | |
| $\sigma^2$ | | | | | | | | | | | | | | | | | | |
| $	au_{00}$ | | | | | | | | | | | | | | | | | | |
| $\tau_{11}$ | | | | | | | | | | | | | | | | | | |
| $\rho_{01}$ | | | | | | | | | | | | | | | | | | |
| ICC | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Observations | | | | | | | | | | | | | | | | | | |
| Marginal R <sup>2</sup> / | | | | | | | | | | _ | | | | | | _ | | |
| Conditional R <sup>2</sup> | | | | | | | | | | | | | | | | | | |
| AIC | | | | | | | | | | | | | | | | | | |

Note—Make ATR the reference group so the estimate tells us how the combined CPS groups compare

Table 6
Best-Fitting Models Predicting Self-Reported Adherence for CPS-T versus CPS-C (N = 23)

| Dependent | VAS | lw | | VAS2w | | | VAS3w | | | VAS1m | | | VAS2m | | | VAS3m | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Variables | | • | | | | | | | | | | | | | | | | |
| | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p | Estimates | CI | p |
| Fixed Effects | | | | | | | | | | | | | | | | | | |
| Intercept | | | | | | | | | | | | | | | | | | |
| Time | | | | | | | | | | | | | | | | | | |
| Intervention | | | | | | | | | | | | | | | | | | |
| Group (CPS-T | | | | | | | | | | | | | | | | | | |
| versus CPS-C) | | | | | | | | | | | | | | | | | | |
| Random Effects | | | | | | | | | | | | | | | | | | |
| $\sigma^2$ | | | | | | | | | | | | | | | | | | |
| $	au_{00}$ | | | | | | | | | | | | | | | | | | |
| $\tau_{11}$ | | | | | | | | | | | | | | | | | | |
| $ ho_{01}$ | | | | | | | | | | | | | | | | | | |
| ICC | | | | | | | | | | | | | | | | | | |
| N | | | | | | | | | | | | | | | | | | |
| Observations | | | | | | | | | | | | | | | | | | |
| Marginal R <sup>2</sup> / | | | | | | | | | | | | | | | | | | |
| Conditional R <sup>2</sup> | | | | | | | | | | | | | | | | | | |
| AIC | | | | | | | | | | | | | | | | | | |

Note—Make CPS-C the reference group so the estimate tells us how CPS-T compares

Table 7
Exploratory Analyses Estimating Effect Sizes Using Self-Reported Outcomes Past Week (Pre-Post... Baseline to 12 weeks)

| Subgroup | n | d | CI | n | Subgroup | n | d | CI | n |
|---|---|---|---|---|---|---|---|---|---|
| VAS1w | rı | и | CI | p | Subgroup | rı | и | CI | p |
| Total Sample | | | | | Young Men | | | | |
| CPS Combined vs. ATR | 34 | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | 54 | | | | CPS-T vs. CPS-C | | | | |
| Sickle Cell Disease | | | | | Young Women | | | | |
| CPS Combined vs. ATR | 14 | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | 1. | | | | CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant | | | | | Latinx | | | | |
| CPS Combined vs. ATR | 10 | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes | | | | | Black | | | | |
| CPS Combined vs. ATR | 10 | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| VAS2w | | | | | | | | | |
| Total Sample $(N = 34)$ | | | | | Young Men | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Sickle Cell Disease $(n = 14)$ | | | | | Young Women | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant $(n = 10)$ | | | | | Latinx | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes $(n = 10)$ | | | | | Black | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| VAS3w | | | | | | | | | |
| Total Sample $(N = 34)$ | | | | | Young Men | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Sickle Cell Disease (n = 14) | | | | | Young Women | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant $(n = 10)$ | | | | | Latinx CDS Combined as ATP | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes ( $n = 10$ )<br>CPS Combined vs. ATR | | | | | Black CDS Combined vs. ATD | | | | |
| | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |

Table 8
Exploratory Analyses Estimating Effect Sizes Using Self-Reported Outcomes Past Month

| Exploratory Analyses Estimating Subgroup | <u>11,1000</u><br>n | $\frac{3i2cs}{d}$ | CI | p | Subgroup | n | d | CI | p |
|---|---|---|---|---|---|---|---|---|---|
| VAS1m | | - | | | <u> </u> | <u> </u> | - | | |
| Total Sample | | | | | Young Men | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Sickle Cell Disease | | | | | Young Women | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant | | | | | Latinx | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes | | | | | Black | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| VAS2m | | | | | Y M | | | | |
| Total Sample | | | | | Young Men | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C<br>Sickle Cell Disease | | | | | CPS-T vs. CPS-C | | | | |
| | | | | | Young Women CPS Combined vs. ATR | | | | |
| CPS Combined vs. ATR<br>CPS-T vs. CPS-C | | | | | CPS Combined vs. ATR CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant | | | | | Latinx | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes | | | | | Black | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| VAS3m | | | | | | | | | |
| Total Sample $(N = 34)$ | | | | | Young Men | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Sickle Cell Disease $(n = 14)$ | | | | | Young Women | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Solid Organ Transplant $(n = 10)$ | | | | | Latinx | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |
| Type 2 Diabetes ( $n = 10$ ) | | | | | Black | | | | |
| CPS Combined vs. ATR | | | | | CPS Combined vs. ATR | | | | |
| CPS-T vs. CPS-C | | | | | CPS-T vs. CPS-C | | | | |